CLINICAL TRIAL: NCT02612090
Title: The Cholesterol Lowering Effects of Strawberry: A Randomized Controlled Trial Establishing Strawberry's Role in Cardiovascular Health
Brief Title: The Cholesterol Lowering Effects of Strawberry
Acronym: STR4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB2015-058
Record Dates: First submitted 2015-11-17; First posted 2015-11-23 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Hypercholesterolemia; Glycemic Response
Keywords: Nutrition; Polyphenols; Berries; Lipid Panels
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Treatment Beverage (Active Comparator): Strawberry
  Interventions: Dietary Supplement: Active Treatment Beverage
- Placebo Treatment Beverage (Placebo Comparator): Placebo Beverage
  Interventions: Dietary Supplement: Placebo Treatment Beverage

INTERVENTIONS:
Dietary Supplement: Active Treatment Beverage — Strawberry
  Other Names: Active Comparator
  Arms: Active Treatment Beverage
Dietary Supplement: Placebo Treatment Beverage — Placebo
  Other Names: Placebo Comparator
  Arms: Placebo Treatment Beverage

SUMMARY:
Primary objective is to assess strawberry intake on LDL cholesterol and its association with atherosclerosis development.

DETAILED DESCRIPTION:
The trial is designed as a randomized, 2-arm, 2-sequence, within-subject, cross-over, chronic feeding study. The arms of the study will include regular consumption of a strawberry or strawberry-placebo powder equivalent to ~3.5 servings of strawberries/day (50g) freeze-dried strawberry powder (provided twice a day, 25 grams each time >6h apart).

A planned sample size of 50 men and women will be enrolled into the study. This study will require one initial screening visit, 4 study visits, and 6 weekly visits. This study will take approximately 12 weeks per subject to complete.

The initial screening visit will provide subject with the informed consent document and determine subject eligibility through anthropometric measurements, vital signs, fasting blood glucose test (finger prick), fasting blood draw, and completion of a survey relate to general eating, health, and exercise habits.

If willing and eligible to participate, a 3-day food record (2 weekdays and 1 weekend day) will be instructed at the Screening Visit and collected before study day 1 to assess subjects' baseline dietary intake pattern. Subjects will be instructed to follow a strictly limited polyphenolic diet for 7 days prior to the study and throughout their participation time, while maintaining their usual diet pattern and physical activity, with counseling by staff investigator and/or Registered Dietitian. A dinner meal will be provided the day before the study visit to control the second meal effect from the food and beverage intake of the night before the study visit.

Subject will arrive at the center in a fasted state for at least 10 hours, well hydrated and rested. Each study visit will require blood draws throughout the visit. After evaluation of subject's health status (via anthropometric, vital sign and blood glucose measurements and in-person interview), a Licensed health care professional will take a fasting blood draw with a butterfly needle. Subjects will be randomized to receive a placebo or treatment beverage based on randomized treatment sequences at 4 study visits. The sequences of receiving the beverage treatments at each visit will be randomly assigned to one of two of following sequences: placebo- treatment beverage or treatment beverage -placebo.

Each study visit will involve blood sample collection at time points 0h (fasting) for assessment of change in plasma lipid and lipoprotein markers. Each study visit will involve a 2 flow mediated dilatation procedure to assess endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* Men and post-menopausal women (without menses for 1 year) with moderate hypercholesterolemia as defined by LDL cholesterol between 115mg/dl-165mg/dl and total cholesterol >160mg/dl preferred but not to exceed 240mg/dl
* 40-69 years of age
* Body Mass Index (BMI) range from 25 to 38.9 kg/m2
* Nonsmoker
* No clinical evidence of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease
* Not taking any medications that would interfere with outcomes of the study, i.e. lipid lowering medications, anti-inflammatory drugs, dietary supplements, etc…
* Able to provide informed consent
* Able to comply and perform the procedures requested by the protocol
* Weight stable: not gained or lost weight +/- 5 kg in previous 3 months

Exclusion Criteria:

* Men and women who smoke
* Past smokers: abstinence for minimum 2 years
* Men and women with known or suspected food intolerance, allergies or hypersensitivity
* Men and women known to have/diagnosed with diabetes mellitus
* Men and women who have fasting blood glucose concentrations > 110mg/dL
* Men and women who have uncontrolled blood pressure >120 mmHg/80 mmHg
* Men and women with documented vascular disease, e.g., heart failure, myocardial infarction, stroke, angina, related surgeries, etc...
* Men and women with cancer other than non-melanoma skin cancer in previous 5 years
* Women who are known to be pregnant or who are intending to become pregnant over the course of the study
* Women who are breast-feeding
* Taking medication or dietary supplements that may interfere with the outcomes of the study; e.g., antioxidant supplement, anti-inflammation, lipid lowering medication, blood pressure lowering medication, etc... Subjects may choose to go off dietary supplements (requires 30 days washout); e.g., fish oil, probiotics, etc...
* Men and women who have donated blood within 3 months of the Screening Visit and blood donors/participants for whom participation in this study will result in having donated more than 1500 milliliters of blood in the previous 12 months.
* Men and women who are vegans
* Substance (alcohol or drug) abuse within the last 2 years
* Excessive coffee and tea consumers (> 4 cups/d) and polyphenol consumers (>2 cups fresh/day
* Men and women who do excessive exercise regularly or athlete
* Unstable weight: gained or lost weight +/- 5 kg in previous 3 months
* Women who are taking unstable dose and brand of hormonal contraceptives and/or stable dose and brand less than 6 months.

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2017-07-16 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Changes in plasma LDL cholesterol in 4-week intervention of strawberries vs control treatment. | 4 weeks
  plasma LDL cholesterol

SECONDARY OUTCOMES:
Changes in endothelial function as measured by Flow Medicated Vasodilation (FMD) in 4-week intervention of strawberries vs control treatment. | 4 weeks
  endothelial function as measured by Flow Medicated Vasodilation (FMD)

OTHER OUTCOMES:
Changes in plasma total cholesterol in 4-week intervention of strawberries vs control treatment. | 4 weeks
  plasma total cholesterol
Changes in plasma HDL cholesterol in 4-week intervention of strawberries vs control treatment. | 4 weeks
  plasma HDL cholesterol
Changes in plasma triglycerides in 4-week intervention of strawberries vs control treatment. | 4 weeks
  plasma triglycerides
Changes in plasma glucose in 4-week intervention of strawberries vs control treatment. | 4 weeks
  plasma glucose
Changes in plasma insulin in 4-week intervention of strawberries vs control treatment. | 4 weeks
  plasma insulin
Changes in plasma C-Reactive Protein in 4-week intervention of strawberries vs control treatment | 4 weeks
  plasma C-Reactive Protein

CONTACTS AND LOCATIONS:
Overall Officials: Britt Britt Burton-Freeman, Ph.D, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang L, Xiao D, Zhang X, Sandhu AK, Chandra P, Kay C, Edirisinghe I, Burton-Freeman B. Strawberry Consumption, Cardiometabolic Risk Factors, and Vascular Function: A Randomized Controlled Trial in Adults with Moderate Hypercholesterolemia. J Nutr. 2021 Jun 1;151(6):1517-1526. doi: 10.1093/jn/nxab034. PMID 33758944